CLINICAL TRIAL: NCT04983238
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial With a Single Arm run-in Period to Evaluate the Safety and Efficacy of Sodium Thiosulfate (BYON5667) Eye Drops to Reduce Ocular Toxicity in Cancer Patients Treated With SYD985
Brief Title: Evaluation of Safety and Efficacy of Sodium Thiosulfate (BYON5667) Eye Drops to Reduce Ocular Toxicity in Cancer Patients Treated With SYD985
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BYON5667.002
Record Dates: First submitted 2021-07-12; First posted 2021-07-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab duocarmazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BYON5667 & SYD985 (Experimental): BYON5667 eye drops should be self-administered daily during waking hours. SYD985, every 3 weeks (Q3W)
  Interventions: Drug: BYON5667 & SYD985
- Placebo & SYD985 (Placebo Comparator): Placebo eye drops should be self-administered daily during waking hours. SYD985, every 3 weeks (Q3W)
  Interventions: Drug: Placebo & SYD985

INTERVENTIONS:
Drug: BYON5667 & SYD985 — Ocular administration: BYON5667, Intravenous administration: SYD985
  Other Names: BYON5667: sodium thiosulfate; SYD985: (vic-)trastuzumab duocarmazine
  Arms: BYON5667 & SYD985
Drug: Placebo & SYD985 — Ocular administration: Placebo, Intravenous administration: SYD985
  Other Names: SYD985: (vic-)trastuzumab duocarmazine
  Arms: Placebo & SYD985

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled trial with a single arm run-in period is to evaluate the safety and efficacy of sodium thiosulfate (BYON5667) eye drops to reduce ocular toxicity in cancer patients treated with the antibody-drug conjugate (ADC) SYD985

DETAILED DESCRIPTION:
This multicenter trial has a single arm run-in period followed by a randomized, placebo-controlled, double-blind comparative part. In the single arm part of the trial, patients with HER2-expressing locally advanced or metastatic solid tumours will be enrolled and treated with the antibody-drug conjugate (ADC) SYD985 once every 3 weeks until disease progression or unacceptable toxicity. All patients will receive concomitant BYON5667 eye drops. When the primary safety and efficacy analysis of the BYON5667 eye drops at Day 63 is favorable, the trial may continue to the comparative part in which patients with locally advanced or metastatic HER2-positive breast cancer will be treated with SYD985. Patients will be randomly assigned (1:1) to receive BYON5667 or placebo eye drops.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female, age ≥18 years at the time of signing first informed consent;
2. Patient with histologically-confirmed, unresectable locally advanced or metastatic cancer with the following restriction:

   Single arm part: patient with solid tumours of any origin (excluding gastric tumours and adenocarcinomas of the gastroesophageal junction) who has progressed on standard therapy or for whom no standard therapy exists; Randomized part: patient with breast cancer who had either progression during or after at least two human epidermal growth factor receptor 2 (HER2)-targeting treatment regimens for locally advanced or metastatic disease, or progression during or after [ado-]trastuzumab emtansine treatment for locally advanced or metastatic disease;
3. HER2 tumour status as determined by a local laboratory using immunohistochemistry (IHC) and/or in situ hybridization (ISH):

   Single arm part: at least IHC 1+; Randomized part: IHC 3+ and/or ISH positive;
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
5. Patient should refrain from wearing any kind of contact lenses during trial treatment;
6. Adequate organ function

Main Exclusion Criteria:

1. Current or previous use of prohibited medication as listed in the protocol
2. History of infusion-related reactions and/or hypersensitivity to trastuzumab containing treatment or excipients of the trial treatments which led to permanent discontinuation of the treatment;
3. History or presence of keratitis;
4. Left ventricular ejection fraction (LVEF) < 50%, or a history of clinically significant decrease in LVEF during previous trastuzumab containing treatment leading to permanent discontinuation of treatment;
5. History or presence of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan;
6. History or presence of clinically significant cardiovascular disease;
7. Severe, uncontrolled systemic disease;
8. Symptomatic brain metastases, brain metastases requiring steroids to manage symptoms, or treatment for brain metastases within 8 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of BYON5667 eye drops by assessing the percentage of patients with SYD985-related ocular adverse events Grade >=1 at Day 63 | 63 days
  Percentage of patients with SYD985-related ocular toxicity Grade ≥1 at Day 63

SECONDARY OUTCOMES:
Ocular toxicity | Day 63 or Day 126
  Percentage of patients with SYD985-related ocular toxicity of different grades at Day 63 or Day 126
Tolerability of BYON5667 eye drops by means of Eye Drop Tolerability questionnaire scores | Up to 2 years
  Tolerability of BYON5667 eye drops Questionnaire includes 5 questions with score of 0 (no discomfort) to 10 (most imaginable discomfort)
National Eye Institute Visual Function Questionnaire (NEI VFQ-25) scores | Up to 2 years
  Self-reported validated questionnaire including 25 questions with scores of 1 to maximum 6, from best/worst to worst/best depending on the question
SYD985-related ocular adverse events (AE) | Up to 2 years
  Time to first SYD985-related ocular AE
Discontinuation due to SYD985-related ocular toxicity | Up to 2 years
  Percentage of patients discontinued due to SYD985-related ocular toxicity
Efficacy of SYD985 by assessing the objective response rate (ORR) | Up to 2 years
  Efficacy of SYD985
Efficacy of SYD985 by assessing the progression-free survival (PFS) | Up to 2 years
  Efficacy of SYD985
Efficacy of SYD985 by assessing the overall survival | Up to 2 years
  Efficacy of SYD985
Safety of SYD985 by assessing incidence and severity of treatment-emergent drug-related adverse events | Up to 2 years
  Safety of SYD985

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mommers, PhD, Study Director — Byondis B.V., The Netherlands
Locations (10):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - UZ Leuven, Leuven
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Hôpital Saint Louis, Paris
- Spain (5):
  - Vall d' Hebron, Barcelona
  - ICO I'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitari Arnau de Vilanova, Lleida
  - START Madrid HU Fundacion Jimenez Diaz, Madrid
  - START Madrid HU HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No